CLINICAL TRIAL: NCT06926868
Title: IZABRIGHT-Breast01: A Randomized, Open-label, Inferentially Seamless Phase 2/3 Study of Izalontamab Brengitecan (BMS-986507) Versus Treatment of Physician's Choice in Patients With Previously Untreated, Locally Advanced, Recurrent Inoperable, or Metastatic Triple-negative Breast Cancer (TNBC) or ER-low, HER2-negative BC Who Are Ineligible for Anti-PD1/PD-L1 Treatment
Brief Title: A Study of Izalontamab Brengitecan Versus Chemotherapy in Participants With Previously Untreated, Locally Advanced, Recurrent Inoperable, or Metastatic Triple-negative Breast Cancer Ineligible for Anti-PD(L)1 Drugs (IZABRIGHT-Breast01)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA244-0008; 2024-519871-24 (Other: EU CTR); U1111-1316-1533 (Other: WHO)
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Breast Neoplasms
Keywords: triple-negative breast cancer; antibody-drug conjugate; ER-low/HER2-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Paclitaxel; Capecitabine; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A1 (Experimental)
  Interventions: Drug: Iza-bren
- Arm A2 (Experimental)
  Interventions: Drug: Iza-bren
- Arm B (Active Comparator)
  Interventions: Drug: Nab-paclitaxel; Drug: Paclitaxel; Drug: Capecitabine; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Iza-bren — Specified dose on specified days
  Other Names: BMS-986507; BL-B01D1; Izalontamab brengitecan
  Arms: Arm A1; Arm A2
Drug: Nab-paclitaxel — Specified dose on specified days
  Arms: Arm B
Drug: Paclitaxel — Specified dose on specified days
  Arms: Arm B
Drug: Capecitabine — Specified dose on specified days
  Arms: Arm B
Drug: Carboplatin — Specified dose on specified days
  Arms: Arm B
Drug: Gemcitabine — Specified dose on specified days
  Arms: Arm B

SUMMARY:
The purpose of this study is to assess the efficacy and safety of iza-bren, a bi-specific antibody-drug conjugate against EGFR and HER3 with a topoisomerase inhibitor payload versus treatment of physician's choice (TPC) (paclitaxel, nab-paclitaxel, carboplatin plus gemcitabine, and capecitabine) for the treatment of first-line metastatic triple-negative breast cancer (TNBC) or estrogen receptor (ER)-low, human epidermal growth factor receptor 2 (HER2)-negative BC patients who are not candidates for anti-PD(L)1 therapy and endocrine therapies.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed and documented locally-advanced, recurrent inoperable, or metastatic TNBC (ER < 1%, PgR < 1%, HER2 IHC 0, 1+, or 2+ with ISH negative for HER2 gene amplification) or ER-low, HER2-negative BC (ER and / or PgR 1% to 10%, HER2 IHC 0, 1+, or 2+ with ISH negative for HER2 gene amplification) per ASCO/CAP criteria, based on the most recently analyzed biopsy or other pathology specimen.
* Patients with recurrent disease must have experienced disease relapse at least 6 months after finishing their last therapy with curative intent.
* Patients with TNBC must be considered ineligible for 1L chemotherapy combination treatment with an anti-PD-1 or an anti-PD-L1 due to either one of the following criteria:

  i) Investigator-determined ineligibility based on PD-L1 negative disease determined and documented prior to trial screening as part of SoC; ii) Has experienced disease relapse between 6 to 12 months after the completion of (neo)adjuvant therapy with an anti-PD(L)1; iii) Has a severe auto-immune disease or other contraindication.
* Patients with ER-low, HER2-negative BC must be ineligible, in the opinion of the Investigator, for endocrine therapy-based treatments.
* No previous systemic therapy in the locally advanced, recurrent inoperable or metastatic setting (ie incurable setting).
* Measurable disease by CT or MRI as per RECIST v1.1.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2028-03-13 (Estimated); Study Completion 2030-05-15 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Approximately 31 months from first participant randomization
  Assessed using Response Evaluation Criteriain Solid Tumors version 1.1 (RECIST v1.1) byblinded independent central review (BICR)

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately up to 57 months from first participant randomization
Recommended Phase 3 Dose (RP3D) of BMS-986507 | Approximately 19 months from first participant randomization
Number of participants with treatment-related Adverse Events (AEs) | Approximately up to 57 months from first participant randomization
Number of participants with laboratory abnormalities | Approximately up to 57 months from first participant randomization
Number of participants with serious AEs (SAEs) | Approximately up to 57 months from first participant randomization
Number of participants with AEs leading to treatment discontinuation, interruption, dose reduction or dose delay | Approximately up to 57 months from first participant randomization
Number of deaths | Approximately up to 57 months from first participant randomization
Objective Response (OR) | Approximately 31 months from first participant randomization
PFS rate | Approximately 19 months from first participant randomization
  Assessed using RECIST v1.1 by BICR
PFS | Approximately 31 months from first participant randomization
  Assessed by Investigator
Disease control rate (DCR) | Approximately 31 months from first participant randomization
Duration of Response (DOR) | Approximately 31 months from first participant randomization
Time to Response (TTR) | Approximately 31 months from first participant randomization
Time to subsequent treatment (TTST) | Approximately up to 57 months from first participant randomization
  Defined as time from randomization to the start of subsequent therapy or death
Progression-free survival after next line of treatment (PFS2) | Approximately up to 57 months from first participant randomization
  Defined as the time from randomization to the date of investigator-defined documented disease progression after next line of treatment or death due to any cause, whichever comes first
Change from baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Approximately up to 57 months from first participant randomization
Change from baseline in EORTC Breast Cancer-specific Quality of Life Questionnaire (QLQ-BR23) | Approximately up to 57 months from first participant randomization
Functional Assessment of Chronic Illness Therapy item GP5 (FACIT GP5) score | Approximately up to 57 months from first participant randomization
Change from baseline in European Quality of Life 5 Dimensions 5 Levels (EQ-5D-5L) | Approximately up to 57 months from first participant randomization
Relative change in tumor size | Approximately up to 19 months from first participant randomization
ORR by RECIST v1.1 per Investigator | Approximately 31 months from first participant randomization

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (292):
- United States (45):
  - Local Institution - 0303, Hot Springs, Arkansas
  - Helios Clinical Research, Cerritos, California
  - Local Institution - 0307, Cerritos, California
  - Local Institution - 0308, Cerritos, California
  - Local Institution - 0309, Cerritos, California
  - Local Institution - 0311, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Local Institution - 0358, Stanford, California
  - Local Institution - 0289, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Local Institution - 0282, Miami, Florida
  - Local Institution - 0296, Pembroke Pines, Florida
  - Local Institution - 0294, Atlanta, Georgia
  - Local Institution - 0357, Atlanta, Georgia
  - Local Institution - 0278, Chicago, Illinois
  - Local Institution - 0280, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Local Institution - 0324, O'Fallon, Illinois
  - Local Institution - 0286, Covington, Louisiana
  - Local Institution - 0288, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - 0359, Detroit, Michigan
  - Minnesota Oncology Hematology, Maple Grove, Minnesota
  - Local Institution - 0372, Minneapolis, Minnesota
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Local Institution - 0312, New York, New York
  - Local Institution - 0279, New York, New York
  - Clinical Research Alliance, Westbury, New York
  - White Plains Hospital, White Plains, New York
  - Local Institution - 0276, Durham, North Carolina
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Local Institution - 0310, Philadelphia, Pennsylvania
  - Local Institution - 0360, Pittsburgh, Pennsylvania
  - St Francis Cancer Center, Greenville, South Carolina
  - Texas Oncology - Central/South Texas, Austin, Texas
  - Texas Oncology - West Texas, El Paso, Texas
  - Texas Oncology - Northeast Texas, Flower Mound, Texas
  - (USOR) Texas Oncology, Houston, Texas
  - Bon Secours St. Francis Medical Center, Midlothian, Virginia
  - Local Institution - 0301, Roanoke, Virginia
  - Shenandoah Oncology, P.C., Winchester, Virginia
- Argentina (10):
  - Local Institution - 0011, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0214, ABB, Buenos Aires F.D.
  - Hospital Italiano de Córdoba, Córdoba, Córdoba Province
  - Centro Privado de RMI Río Cuarto S.A. II, Río Cuarto, Córdoba Province
  - Sanatorio Plaza, Rosario, Santa Fe Province
  - Instituto Argentino de Diagnóstico y Tratamiento (IADT), Buenos Aires
  - Centro Oncologico Korben, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Local Institution - 0346, Buenos Aires
  - Local Institution - 0348, Mendoza
- Australia (6):
  - Local Institution - 0170, Macquarie University, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Grampians Health, Ballarat Central, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - St. John of God Subiaco Hospital, Subiaco, Western Australia
- Austria (5):
  - Medizinische Universität Graz, Graz, Styria
  - Medizinische Universitaet Innsbruck, Innsbruck, Tyrol
  - Uniklinikum Salzburg, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien, Vienna
- Brazil (10):
  - Local Institution - 0187, Manaus, Amazonas
  - Local Institution - 0147, Fortaleza, Ceará
  - CEDOES, Vitória, Espírito Santo
  - Local Institution - 0159, Curitiba, Paraná
  - Futtura Oncology - Clinical Research Hub, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Local Institution - 0164, São José do Rio Preto, São Paulo
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro
  - Clínica de Pesquisas e Centro de Estudos em Oncologia Ginecológica e Mamária Ltda, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo
- Canada (7):
  - BC Cancer Kelowna, Kelowna, British Columbia
  - Local Institution - 0217, Victoria, British Columbia
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Intégré de Santé et de Services Sociaux de Lanaudière, Saint-Charles-Borromée, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke (CIUS, Sherbrooke, Quebec
- Chile (5):
  - Local Institution - 0016, Viña del Mar, Región de Valparaíso
  - Local Institution - 0138, Santiago, Santiago Metropolitan
  - Local Institution - 0021, Santiago, Santiago Metropolitan
  - Local Institution - 0017, Santiago, Santiago Metropolitan
  - Local Institution - 0018, Santiago, Santiago Metropolitan
- China (30):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Local Institution - 1005, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, BEI
  - Local Institution - 1006, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fyzhou, Fujian
  - Local Institution - 1016, Xiamen, Fujian
  - Local Institution - 1031, Lanzhou, Gansu
  - Guangxi Medical University Affiliated Cancer Hospital, Nanning, Guangxi
  - Local Institution - 1028, Harbin, Harbin
  - Anyang Cancer Hospital, Anyang, Henan
  - Local Institution - 1009, Zhengzhou, Henan
  - Local Institution - 1032, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Local Institution - 1011, Changsha, HUN
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Local Institution - 1012, Changchun, Liaoning
  - Local Institution - 1014, Shenyang, Liaoning
  - Local Institution - 1017, Jinan, Shandong
  - Local Institution - 1015, Qingdao, Shandong
  - Local Institution - 1018, Taiyuan, Shanxi
  - Sichuan Provincial People'S Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Local Institution - 1020, Tianjin, Tianjin Municipality
  - Local Institution - 1029, Kunming, Yunnan
  - Local Institution - 1023, Hangzhou, Zhejiang
  - Local Institution - 1025, Guangzhou
- Colombia (8):
  - Local Institution - 0195, Medellín, Antioquia
  - Local Institution - 0201, Rionegro, Antioquia
  - Local Institution - 0194, Barranquilla, Atlántico
  - Local Institution - 0182, Puerto Colombia, Atlántico
  - Local Institution - 0181, Montería, COR
  - Local Institution - 0327, Bogota, Cundinamarca
  - Local Institution - 0183, Cali, Valle del Cauca Department
  - Local Institution - 0349, Medellín
- France (13):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - Local Institution - 0090, Lyon, Auvergne-Rhône-Alpes
  - Local Institution - 0272, Dijon, Côte-d'Or
  - Local Institution - 0098, Toulouse, Haute-Garonne
  - Institut Régional du Cancer Montpellier, Montpellier, Hérault
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer, Rennes, Ille-et-Vilaine
  - Local Institution - 0092, Saint-Herblain, Loire-Atlantique
  - Local Institution - 0091, Reims, Marne
  - Gustave Roussy, Villejuif, Paris
  - Institut Paoli-Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
  - Local Institution - 0096, Clermont-Ferrand, Puy-de-Dôme
  - Centre Oscar Lambret, Lille
  - Local Institution - 0088, Paris
- Germany (16):
  - Klinikum Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Klinikum Augsburg, Augsburg, Bavaria
  - Rotkreuzklinikum München gemeinnützige GmbH, München, Bavaria
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt am Main, Hesse
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Langen, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Luisenkrankenhaus Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung, Essen, North Rhine-Westphalia
  - Local Institution - 0254, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Charité - Universitaetsmedizin Berlin - Campus Bejnamin Franklin, Berlin
  - Vivantes Klinikum Am Urban, Berlin
  - Gynaekologisches Zentrum Bonn, Bonn
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Ulm, Ulm
- Greece (4):
  - Local Institution - 0043, Athens, Attikí (Region)
  - Agios Savvas Regional Cancer Hospital, Athens, Attikí
  - Local Institution - 0038, Athens, Attikí
  - Local Institution - 0086, Heraklion, Irakleío
- India (9):
  - Local Institution - 0337, Mumbai, Maharashtra
  - Local Institution - 0131, Mumbai, Maharashtra
  - Local Institution - 0134, Nagpur, Maharashtra
  - Local Institution - 0352, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0266, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0206, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0125, Chennai, Tamil Nadu
  - Local Institution - 0130, Hyderabad, Telangana
  - Local Institution - 0133, Varanasi, Uttar Pradesh
- Israel (5):
  - Local Institution - 0186, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Hillel Yaffe Medical Center, Hadera, Northern District
  - Rambam Health Care Campus, Haifa, Northern District
- Italy (11):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli, Campania
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna, Emilia-Romagna
  - Cro-Irccs, Aviano, Friuli Venezia Giulia
  - Ospedale San Martino, Genoa, Liguria
  - Ospedale "Felice Lotti" Di Pontedera, Pontedera, Pisa
  - Nuovo Ospedale di Prato-S.Stefano, Prato, Tuscany
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Local Institution - 0058, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - Local Institution - 0056, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
- Japan (25):
  - Local Institution - 0236, Nagoya, Aichi-ken
  - Local Institution - 0230, Chiba, Chiba
  - Local Institution - 0240, Matsuyama, Ehime
  - Local Institution - 0226, Otashi, Gunma
  - Local Institution - 0222, Sapporo, Hokkaido
  - Local Institution - 0232, Kanazawa, Ishikawa-ken
  - Local Institution - 0234, Isehara, Kanagawa
  - Local Institution - 0237, Yokohama, Kanagawa
  - Local Institution - 0246, Tsu, Mie-ken
  - Local Institution - 0223, Sendai, Miyagi
  - Local Institution - 0238, Suita, Osaka
  - Local Institution - 0227, Hidaka, Saitama
  - Local Institution - 0224, Ina-machi, Saitama
  - Local Institution - 0231, Bunkyo-ku, Tokyo
  - Local Institution - 0229, Chuo-ku, Tokyo
  - Local Institution - 0228, Koto, Tokyo
  - Local Institution - 0245, Shinagawa, Tokyo
  - Local Institution - 0233, Shinjuku-ku, Tokyo
  - Local Institution - 0242, Fukuoka
  - Local Institution - 0225, Fukushima
  - Local Institution - 0243, Hiroshima
  - Local Institution - 0244, Kagoshima
  - Local Institution - 0235, Kyoto
  - Local Institution - 0241, Okayama
  - Local Institution - 0239, Osaka
- Mexico (10):
  - Local Institution - 0177, Mexico City, DIF
  - Local Institution - 0264, Tijuana, Estado de Baja California
  - Local Institution - 0178, Guadalajara, Jalisco
  - Local Institution - 0329, Mexico City, Mexico City
  - Local Institution - 0175, Monterrey, Nuevo León
  - Local Institution - 0176, Monterrey, Nuevo León
  - Local Institution - 0355, Monterrey, Nuevo León
  - Local Institution - 0173, Oaxaca City, Oaxaca
  - Local Institution - 0179, Mérida, Yucatán
  - Local Institution - 0174, Chihuahua City
- Poland (6):
  - Local Institution - 0189, Skórzewo, Greater Poland Voivodeship
  - Local Institution - 0074, Biała Podlaska, Lublin Voivodeship
  - Local Institution - 0072, Warsaw, Masovian Voivodeship
  - Mazowiecki Szpital Onkologiczny, Warsaw, Masovian Voivodeship
  - Local Institution - 0076, Opole, Opole Voivodeship
  - Local Institution - 0221, Lodz, Łódź Voivodeship
- Portugal (7):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, Lisbon, Lisbon District
  - Local Institution - 0106, Lisbon, Lisbon District
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon, Lisbon District
  - Local Institution - 0124, Coimbra
  - Hospital da Luz Lisboa, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Local Institution - 0253, Porto
- Romania (11):
  - Local Institution - 0212, Bistriţa, Bistrița-Năsăud County
  - Local Institution - 0213, Bucharest, București
  - SC Radiotherapy Center Cluj SRL, Florești, Cluj
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Local Institution - 0084, Ploieşti, Prahova
  - Cabinet Medical Oncomed, Timișoara, Timiș County
  - Spitalul Clinic Filantropia, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Centrul de Radioterapie Amethyst Timis, Dumbrăviţa
  - S.C. Centrul de Oncologie Euroclinic S.R.L., Iași
  - Institutul Regional de Oncologie, Iași
- South Africa (6):
  - Local Institution - 0351, East London, Eastern Cape
  - Local Institution - 0342, Parktown, Gauteng
  - Local Institution - 0336, Pretoria, Gauteng
  - Local Institution - 0341, Pretoria, Gauteng
  - Local Institution - 0340, Soweto, Gauteng
  - Local Institution - 1034, Panorama, Western Cape
- South Korea (8):
  - Local Institution - 0066, Goyang-si, Kyǒnggi-do
  - Local Institution - 0067, Seongnam, Kyǒnggi-do
  - Local Institution - 0068, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0063, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0071, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0064, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0065, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0069, Daegu, Taegu-Kwangyǒkshi
- Spain (12):
  - CHUAC-Hospital Teresa Herrera, A Coruña, A Coruña [La Coruña]
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0172, Hospitalet, Barcelona [Barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Beata María Ana, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- Sweden (5):
  - Skånes Universitetssjukhus Malmö, Malmo, Skåne Län [se-12]
  - Local Institution - 0026, Stockholm, Stockholms Län [se-01]
  - Akademiska sjukhuset, Uppsala, Uppsala Län [se-03]
  - Universitetssjukhuset Örebro, Örebro, Örebro Län [se-18]
  - Universitetssjukhuset i Linköping, Linköping, Östergötlands Län [se-05]
- Switzerland (3):
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - CHUV (centre hospitalier universitaire vaudois), Lausanne, Canton of Vaud
  - Brust-Zentrum, Zurich
- Turkey (Türkiye) (4):
  - Local Institution - 0361, Adana
  - Local Institution - 0362, Ankara
  - Local Institution - 0364, Istanbul
  - Local Institution - 0363, Istanbul
- United Arab Emirates (4):
  - Local Institution - 0323, Abu Dhabi, Abu Dhabi Emirate
  - Local Institution - 0318, Abu Dhabi, Abu Dhabi Emirate
  - Local Institution - 0322, Al Ain City, Abu Dhabi Emirate
  - Local Institution - 0319, Abu Dhabi
- United Kingdom (7):
  - The Royal Cornwall Hospital, Truro, England
  - St Bartholomew's Hospital, London, London, City of
  - Guy's & St Thomas' NHS Foundation Trust, London, London, City of
  - Local Institution - 0204, London, London, City of
  - Local Institution - 0171, Belfast
  - The Christie NHS Foundation Trust, Manchester
  - Local Institution - 0006, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06926868.html